CLINICAL TRIAL: NCT06198413
Title: A Dose-Escalation Study of LX102 Gene Therapy for Neovascular Age-Related Macular Degeneration (nAMD)
Brief Title: LX102 in Patients With Neovascular Age-Related Macular Degeneration (nAMD)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Innostellar Biotherapeutics Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INNOSTELLAR-LX102A01-1
Record Dates: First submitted 2023-12-25; First posted 2024-01-10 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Neovascular Age-Related Macular Degeneration
Keywords: Age-related macular degeneration; AMD; Neovascular AMD; Neovascular age-related macular degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- LX102 Dose 1 (Experimental): Low dose of LX102
  Interventions: Genetic: LX102 subretinal injection
- LX102 Dose 2 (Experimental): Mid dose of LX102
  Interventions: Genetic: LX102 subretinal injection
- LX102 Dose 3 (Experimental): High dose of LX102
  Interventions: Genetic: LX102 subretinal injection

INTERVENTIONS:
Genetic: LX102 subretinal injection — LX102: AAV-based gene therapy comprised of codon-optimized sequence encoding VEGF-trap

SUMMARY:
The goal of this study is to evaluate the safety and efficacy of LX102 gene therapy for nAMD.

DETAILED DESCRIPTION:
This study will enroll subjects aged ≥ 50 years old to receive a single unilateral subretinal injection of LX102 to evaluate its safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign the informed consent, and willing to attend follow-up visits.
2. Age ≥ 50
3. Diagnosis of active CNV secondary to neovascular AMD
4. BCVA ETDRS letters between 5 and 63
5. Subjects must have received a minimum of 2 injections within 6 months prior to screening
6. Demonstrated a meaningful response to anti-VEGF therapy

Exclusion Criteria:

1. CNV or macular edema in the study eye secondary to diseases other than nAMD
2. Retinal detachment, uveitis, uncontrolled glaucoma in the study eye, or any condition preventing visual acuity improvement
3. Acute coronary syndrome, myocardial infarction or coronary artery revascularization, CVA, TIA in the last 6 months
4. Uncontrolled hypertension defined as average SBP ≥160 mmHg or an average DBP ≥100 mmHg
5. Uncontrolled diabetes defined as HbA1c >7.5%

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) | 4 weeks
  Incidence of dose-limiting toxicity (DLT) following LX102 subretinal injection at different doses
Incidence of adverse events (AEs) and serious adverse events (SAEs) | 52 weeks
  Incidence of ocular and systemic adverse events (AEs) and serious adverse events (SAEs) following LX102 subretinal injection

SECONDARY OUTCOMES:
Mean change in BCVA from Baseline | 12 weeks, 36 weeks 52 weeks
  BCVA measured by ETDRS
Mean change in Central Subfield Thickness (CST) from Baseline | 12 weeks, 36 weeks 52 weeks
  CST measured by spectral domain optical coherence tomography (SD-OCT)
Mean time from LX102 administration to anti-VEGF rescue injection for the first time | 52 weeks
Percentage of participants requiring anti-VEGF rescue injection | 52 weeks
Mean number of anti-VEGF rescue injections | 52 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Zhejiang University Eye Hospital, Hangzhou, Zhejiang
  - Shanghai General Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No